CLINICAL TRIAL: NCT04355689
Title: Safety and Efficacy of NPI-001 Tablets Versus Placebo for Treatment of Retinitis Pigmentosa Associated With Usher Syndrome
Brief Title: Safety and Efficacy of NPI-001 Tablets for RP Associated With Usher Syndrome
Acronym: SLO RP
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nacuity Pharmaceuticals, Inc. (Industry)
Collaborators: Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-18-04
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Usher Syndromes
Keywords: retinitis pigmentosa Usher vision NPI-001 tablet
MeSH Terms: conditions — Usher Syndromes

STUDY DESIGN:
Intervention Model Description: NPI-001 Tablets versus Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPI-001 (Experimental): NPI-001 Tablet, 250 mg, BID
  Interventions: Drug: NPI-001
- Placebo (Placebo Comparator): Placebo Tablet, BID
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NPI-001 — oral tablet
  Arms: NPI-001
Other: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
This study will examine the safety and efficacy of NPI-001 Tablets as compared to placebo for 24 months in subjects with vision loss due to RP associated with Usher syndrome.

DETAILED DESCRIPTION:
This study will examine the safety and efficacy of oral NPI-001 Tablets as compared to oral placebo tablets for 24 months in subjects with vision loss due to RP associated with Usher syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years.
2. Able to comprehend and willing to sign an informed consent form (ICF) and to adhere to the study protocol.
3. Diagnosed with Usher syndrome.
4. EZ zone with width ≥500 microns, which includes the fovea in each eye at Visit 2, (Screen B).
5. Have at least 20 detectable points on the MAIA grid.
6. On stable dose of medications associated with other conditions for at least one month.
7. Both female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a bilateral oophorectomy, hysterectomy or bilateral salpingectomy; must abstain from intercourse; or must agree to practice 2 acceptable methods of contraception throughout the course of the study and 4 weeks after the last visit. Acceptable methods of contraception include hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring), intrauterine device, barrier methods (diaphragm, condom) with spermicide, tubal ligation, or vasectomy.

Exclusion Criteria:

Ocular:

1. All edges of the EZ area in both eyes cannot be visualized at Visit 2 (Screen B).
2. Concurrent retinal pathologies that result in vision loss or inability to fixate, including but not limited to, choroideremia, retinal vein occlusion, and neovascular age-related macular degeneration.
3. Intraocular surgery within the last two months or capsulotomy within the last month.
4. History of uveitis, Coat's disease, diabetic retinopathy, glaucoma, herpes simplex of the eye, or currently has a cataract that prevents visualization of the posterior pole.
5. Unstable fixation during microperimetry in either eye at either screening or baseline visits.

   Non-Ocular:
6. Use of any other investigational new drug, or participation in another clinical trial within 12 weeks before the start of study treatment.
7. Use of N-acetylcysteine containing products in the previous 30 days prior to the baseline visit or unwilling to refrain from such supplements for the duration of the study.
8. Liver or kidney disease, cystic fibrosis, asthma or chronic obstructive pulmonary disease (COPD), history of thrombocytopenia not due to a reversible cause, or other blood dyscrasia.
9. Suspected liver dysfunction determined by having alanine aminotransferase (ALT), aspartate aminotransferase (AST), or bilirubin values > 1.5 X the upper limit of normal (ULN).
10. Platelet or hemoglobin values that are below the lower limit of normal at screening (subjects with normal hemoglobin and mean corpuscular volume below the lower limit of normal should have iron studies performed to ensure that they are iron replete before taking part in the study), or neutrophils or white cell count which is above the upper limit of normal.
11. Presence of more than + proteinuria on urinalysis at screening or (confirmed by abnormal albumin creatinine ratio).
12. Presence of hematuria on urinalysis at screening. (If hematuria is detected on urinalysis, then the specimen should be subjected to microscopy, and subject should be excluded if more than 10 X 106 red blood cells/L.) If the subject is a female in whom the hematuria may be due to menses, then the urinalysis can be repeated after a few days.
13. C-reactive protein (CRP) value above 10 mg/L.
14. Subject has a recent history of presence of gross blood in stools.
15. History of known sensitivity to N-acetylcysteine or similar thiol compounds.
16. History of hypersensitivity to any medication or food resulting in systemic symptoms.
17. History of cancer (other than non-melanoma skin cancer) diagnosed or requiring treatment within the past 2 years.
18. Pregnant women or women planning to become pregnant in the next 25 months or men with partners planning to become pregnant in the next 25 months.
19. Lactating women who are breast-feeding.
20. A potential participant lives in the same household as a current participant in this study.
21. Inability to provide blood samples, including difficulty with venous access.
22. Any reason, in the opinion of the Principal Investigator, the subject should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate change from baseline for retinal sensitivity assessed by microperimetry of active versus placebo | 24 months
  Evaluate change from baseline for retinal sensitivity assessed by microperimetry of active versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Lee Anderson, MD, Study Chair — Nacuity Pharmaceuticals, Inc.
Locations (4):
- Australia (4):
  - Queensland Eye Institute, Brisbane
  - CERA, Melbourne
  - Lions Eye Institute, Perth
  - Sydney Eye Hospital / Save Sight Institute, Sydney

IPD SHARING:
Plan to Share IPD: No